CLINICAL TRIAL: NCT00372411
Title: CSP #558 - Robotic Assisted Upper-Limb Neurorehabilitation in Stroke Patients
Brief Title: Robotic Assisted Upper-Limb Neurorehabilitation in Stroke Patients
Acronym: VA ROBOTICS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Burke Medical Research Institute (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 558
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Single-blind; Clinical Trial; Randomized controlled trial; Upper extremity; Robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Robot-Assisted Therapy - MIT-MANUS System
  Interventions: Device: Robot-Assisted Therapy - MIT-MANUS System
- Arm 2 (Active Comparator): Intensive Comparison Therapy
  Interventions: Other: Intensive Comparison Therapy
- Arm 3 (Other): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Robot-Assisted Therapy - MIT-MANUS System — The MIT-MANUS robot consists of four modules to train the entire upper limb: module A: shoulder-elbow; module B: anti-gravity; module C: wrist, and module D: hand-unit. Training will be given for 12 weeks and is divided into 4 consecutive blocks, with 9 training sessions per block.
  Arms: Arm 1
Other: Intensive Comparison Therapy — The intensive comparison therapy protocol being used in CSP#558 was developed and field-tested at the Burke Rehabilitation Hospital. It exposes the patient to the identical number of treatments, time, and intensity that robot treated patients will receive (12 weeks, 3 times per week). Therapy sessions can be conducted on back-to-back days if needed and on more than 3 days a week (with approval from the Study Chairman) over a treatment period of up to 14 weeks in order to complete the 36 treatment sessions. During each 1-hour session, subjects participate in therapy in four successive stages: 1) warm-up and assisted stretching; 2) active arm treatments; 3) goal-directed planar reaching, and 4) functionally based Neurodevelopment Techniques (NDT)/Bobath arm training (Bobath, 1979).
  Other Names: ICT
  Arms: Arm 2
Other: Usual Care — The usual chronic stroke care as delivered at each participating medical center
  Arms: Arm 3

SUMMARY:
This study will compare robotic training with usual care and intensive comparison therapy to attempt to improve upper extremity function.

DETAILED DESCRIPTION:
Primary Hypothesis: The primary hypothesis is that robotic training compared with usual care and intensive comparison therapy will lead to improved upper extremity function. Eligible patients will be randomized to one of three treatment arms: 1) usual care, 2) intensive comparison therapy, or 3) robotic training. Participants assigned to intensive comparison therapy or robot-assisted training will receive treatment for 12 weeks consisting of three one-hour sessions a week and then usual care for the remainder of follow-up. Those assigned to usual care will receive the usual stroke care as delivered at each participating medical center for 36 weeks and then will be offered, as compassionate care, their choice of either robot-assisted or intensive comparison therapy.

Secondary Hypothesis: The secondary hypotheses are that compared with usual care and intensive comparison therapy, robotic treatment will lead to improved quality of life and task performance involving proximal and distal control of the paretic arm. If the robotic arm is effective, two other secondary objects are to evaluate its early (less than 12 week) and late (36 week) effects on the primary and secondary outcomes.

Primary Outcome: The primary study outcome is the change in the Fugl-Meyer score of neurological impairment at 12 weeks relative to baseline.

Secondary Outcome: Secondary outcomes include the Stroke Impact Scale and Wolf Motor Function Test. A cost-effectiveness analysis is planned but only will be conducted if robotic training is more effective than usual care.

Study Abstract: CSP #558 will be a randomized, multi-center, outpatient phase II trial to assess the safety and efficacy of robot-assisted therapy for neurorehabilitation in stroke patients with moderate to severe upper extremity impairment.

The target sample is 158 patients: 26 usual care, 66 intensive comparison therapy and 66 robot training. This sample size will provide 90% power to detect a 5-point mean difference in the Fugl-Meyer scale between robot training and usual care and 3-point mean difference between robot training and intensive comparison therapy. There will be one interim analysis of the primary endpoint at 12 months for the purpose of sample size re-estimation using an adaptive design. The planned study duration is 33 months with 24 months of intake and nine months of follow-up.

IMPACT STATEMENT

If robotic training proves to be beneficial it will not only provide a functionally-oriented and neurophysiologically appropriate therapy, but also will make more widely available high-quality, evidence-based rehabilitative care at a time when there is a shortage of experienced therapists and a progressively growing rehabilitative need for veterans and all Americans.

ELIGIBILITY:
Inclusion Criteria:

* A single new focal unilateral stroke with diagnosis verified by brain imaging (MRI) or CT scan that has occurred at least 6 months prior to enrollment.
* Age 18 years of age and older.
* Upper extremity Fugl-Meyer score >=7 or <=38 (max 66). (These thresholds include neither hemiplegic nor fully recovered motor function in 14 muscles of the shoulder, elbow, and wrist.)
* Cognitive function sufficient to understand the experiments and follow instructions (Mini-Mental Status Score of 22 and higher or interview for aphasic subjects).
* Willingness to avoid any new alternative arm rehabilitative approaches for the duration of the study.
* Written informed consent to participate in the study.

Exclusion Criteria:

* A fixed contracture in the affected limb that prevents movement along the entire dynamic range required by either robot-assisted or intensive comparison therapy.
* Joint pain that occurs within the range of motion required by the intervention protocols (intensive comparison therapy and robot-assisted therapy).
* Enrolled in or planning to enroll in another interventional research trial that involves the upper limbs using procedures proposed to enhance or limit the function of the upper extremity (such as adjuvant rehabilitation or Botox injections) during the 36 weeks of participation.
* Prior experience with robot-assisted therapy or intensive comparison therapy for the upper limb as described in this specific study.
* A complicating medical condition that would prevent completion of the trial.
* Unable to complete the nine-month study, e.g., extended planned vacation.
* Any other known pre-existing bone diseases that might increase the risk of bone fracture or other injury from intensive comparison therapy or robot-assisted therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-12; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, MD PhD, Study Chair — Providence VA Medical Center
Locations (5):
- United States (5):
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - Providence VA Medical Center, Providence, Rhode Island
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Result] Lo AC, Guarino P, Krebs HI, Volpe BT, Bever CT, Duncan PW, Ringer RJ, Wagner TH, Richards LG, Bravata DM, Haselkorn JK, Wittenberg GF, Federman DG, Corn BH, Maffucci AD, Peduzzi P. Multicenter randomized trial of robot-assisted rehabilitation for chronic stroke: methods and entry characteristics for VA ROBOTICS. Neurorehabil Neural Repair. 2009 Oct;23(8):775-83. doi: 10.1177/1545968309338195. Epub 2009 Jun 18. PMID 19541917
- [Result] Lo AC, Guarino PD, Richards LG, Haselkorn JK, Wittenberg GF, Federman DG, Ringer RJ, Wagner TH, Krebs HI, Volpe BT, Bever CT Jr, Bravata DM, Duncan PW, Corn BH, Maffucci AD, Nadeau SE, Conroy SS, Powell JM, Huang GD, Peduzzi P. Robot-assisted therapy for long-term upper-limb impairment after stroke. N Engl J Med. 2010 May 13;362(19):1772-83. doi: 10.1056/NEJMoa0911341. Epub 2010 Apr 16. PMID 20400552
- [Result] Wagner TH, Lo AC, Peduzzi P, Bravata DM, Huang GD, Krebs HI, Ringer RJ, Federman DG, Richards LG, Haselkorn JK, Wittenberg GF, Volpe BT, Bever CT, Duncan PW, Siroka A, Guarino PD. An economic analysis of robot-assisted therapy for long-term upper-limb impairment after stroke. Stroke. 2011 Sep;42(9):2630-2. doi: 10.1161/STROKEAHA.110.606442. Epub 2011 Jul 14. PMID 21757677
- [Derived] Wittenberg GF, Richards LG, Jones-Lush LM, Roys SR, Gullapalli RP, Yang S, Guarino PD, Lo AC. Predictors and brain connectivity changes associated with arm motor function improvement from intensive practice in chronic stroke. F1000Res. 2016 Aug 31;5:2119. doi: 10.12688/f1000research.8603.2. eCollection 2016. PMID 28357039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 11-8-06 and 10-31-08, 200 were screened and 127 randomized from 4 VA medical centers: Gainesville, West Haven, Baltimore, and Seattle. Usual care enrollment was stopped after 15 months when target information was attained per protocol. Recruitment to the robot-assisted and intensive comparison groups continued for 24 months.
Groups:
- Robot-assisted Therapy: Robot-Assisted Therapy uses the MIT-MANUS robot and consists of four modules, shoulder-elbow, anti-gravity, wrist, and hand-unit to train the entire upper limb. Training was given for 12 weeks and was divided into 4 consecutive blocks, with 9 training sessions per block.
- Intensive Comparison Therapy: Intensive comparison therapy consisted of the identical number of treatments, time, and intensity of Robot-assisted therapy (12 weeks, 3 times per week). Each 1-hour therapy session consisted of four successive stages: 1) warm-up and assisted stretching; 2) active arm treatments; 3) goal-directed planar reaching, and 4) functionally based Neurodevelopment Techniques/Bobath arm training.
- Usual Care: Usual Care consisted of the usual chronic stroke care as delivered at each participating medical center.
Period: Overall Study
Arm/Group | Robot-assisted Therapy | Intensive Comparison Therapy | Usual Care
Started | 49 | 50 | 28
Completed | 44 | 42 | 25
Not Completed | 5 | 8 | 3
Not completed — Withdrawal by Subject | 3 | 4 | 1
Not completed — Death | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robot-assisted Therapy | Intensive Comparison Therapy | Usual Care | Total
Number analyzed (Participants) | 49 | 50 | 28 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11) | 64 (11) | 63 (12) | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 47 | 48 | 27 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 48 | 48 | 28 | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 12 | 5 | 27
  White | 38 | 35 | 23 | 96
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 28 | 127
Index Stroke Type [Number; unit: participants]
  Hemorrhagic | 7 | 6 | 6 | 19
  Ischemic | 42 | 44 | 22 | 108
Index Stroke Location [Number; unit: Participants]
  Anterior circulation ≥1/3 of hemisphere | 6 | 14 | 6 | 26
  Anterior circulation <1/3 of hemisphere | 17 | 21 | 10 | 48
  Small deep infarct | 17 | 15 | 6 | 38
  Posterior circulation | 9 | 0 | 6 | 15
Time from Index Stroke to Randomization [Mean (Standard Deviation); unit: Years] | 3.6 (4.0) | 4.8 (4.0) | 6.2 (5.0) | 4.7 (4.2)
Fugl-Meyer Assessment [Mean (Standard Deviation); unit: units on a scale] — Primary outcome baseline scores
  units on a scale | 19.7 (10.7) | 17.3 (8.4) | 20.3 (9.0) | 18.9 (9.5)
Comorbidity Disease Index [Number; unit: participants] — The Comorbidity Disease Index domains include cardiac, respiratory, neurologic, musculoskeletal, general (mental or emotional problems and sleep or pain disorders), cancer, diabetes, and visual problems. The domain scores are totaled to create an overall comorbidity score (≤1, 2, or ≥3 domains).
  participants
    ≤1 Domain | 7 | 7 | 2 | 16
    2 Domains | 13 | 24 | 8 | 45
    ≥3 Domains | 29 | 19 | 18 | 66

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment for Motor Recovery (FM) Scale
Description: Fugl-Meyer (FM) is a standard instrument for the quantitative clinical assessment of motor impairment and function. In this study the upper extremity subsection of the FM was used. The FM assesses several impairment dimensions by using a 3 point ordinal scale: 0 = cannot perform, 1 = can perform partially and 2 = can perform fully. These measures are summed to an overall score is Scoring for upper extremity FM ranges from 0 (worst, completely plegic) to 66 (best, normal). Higher scores indicate better functioning. Outcome measure is the change in the FM score at 6, 12, 24 and 36 weeks relative to baseline.
Time Frame: 6, 12, 24 and 36 weeks minus baseline
Population: All participants with baseline and follow-up measures were included by intention-to-treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Robot-assisted Therapy | Intensive Comparison Therapy | Usual Care
Number analyzed (Participants) | 47 | 46 | 27
units on a scale
  6 weeks minus baseline | 3.01 (0.92) | 3.19 (0.91) | -2.08 (1.08)
  12 weeks minus baseline | 3.87 (1.05) | 4.01 (1.06) | -1.06 (1.00)
  24 weeks minus baseline | 4.22 (1.05) | 2.75 (1.06) | -2.02 (1.14)
  36 weeks minus baseline | 5.07 (1.18) | 2.81 (1.18) | -0.53 (1.19)
Statistical Analysis 1: Comparison: Robot-assisted Therapy vs Usual Care; Because randomization to usual care was stopped after 15 months as specified by the protocol, comparisons of robot-assisted therapy with usual care included only patients who were recruited during this period; Test type: Superiority or Other; p = 0.08, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; Analysis is of change at 12 weeks minus baseline adjusted for the study site as a fixed effect, the Comorbidity Disease Index, and baseline FM value; Mean Difference (Net) = 2.17, 95% CI 2-sided [-0.23 to 4.58]
Statistical Analysis 2: Comparison: Robot-assisted Therapy vs Usual Care; Because randomization to usual care was stopped after 15 months as specified by the protocol comparisons of robot-assisted therapy with usual care included only patients who were recruited during this period; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; Secondary analysis used longitudinal methods to assess the effect of treatment on outcomes over 36 weeks with visits at 6, 12, 24, and 36 weeks; Mean Difference (Net) = 2.88, 95% CI 2-sided [0.57 to 5.18]
Statistical Analysis 3: Comparison: Robot-assisted Therapy vs Intensive Comparison Therapy; Comparisons between robot-assisted therapy and intensive comparison therapy included all patients who underwent randomization and were evaluated; Test type: Superiority or Other; p = 0.92, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.14, 95% CI 2-sided [-2.94 to 2.65]
Statistical Analysis 4: Comparison: Robot-assisted Therapy vs Intensive Comparison Therapy; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.63, Mixed Models Analysis — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 1, analysis 2]; Median Difference (Net) = -0.58, 95% CI 2-sided [-2.97 to 1.81]

2. Secondary Outcome: Stroke Impact Scale
Description: The Stroke Impact Scale (SIS) is stroke specific, self-reported measure that evaluates function and quality of life in eight clinically relevant domains. The domains of hand function, activities of daily living, instrumental activities of daily living, mobility, and social participation were used; total score ranges from 0 to 100 with higher values indicating better functioning. Outcome is change at 6, 12, 24 and 36 weeks relative to baseline.
Time Frame: 6, 12, 24 and 36 weeks minus baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Robot-assisted Therapy | Intensive Comparison Therapy | Usual Care
Number analyzed (Participants) | 47 | 46 | 27
units on a scale
  6 weeks minus baseline | 5.49 (1.61) | 4.08 (1.57) | -3.79 (2.47)
  12 weeks minus baseline | 6.31 (1.68) | 5.77 (1.67) | -3.03 (2.34)
  24 weeks minus baseline | 5.58 (1.68) | 4.23 (1.69) | -0.26 (2.37)
  36 weeks minus baseline | 5.14 (1.89) | 4.97 (1.88) | 0.76 (2.49)
Statistical Analysis 1: Comparison: Robot-assisted Therapy vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.009, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; Analysis is change at 12 weeks minus baseline, adjusted for study site as a fixed effect, Comorbidity Disease Index, and the baseline SIS value; Mean Difference (Net) = 7.64, 95% CI 2-sided [2.03 to 13.24]
Statistical Analysis 2: Comparison: Robot-assisted Therapy vs Usual Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 1, analysis 2]; Mean Difference (Net) = 5.95, 95% CI 2-sided [0.34 to 11.56]
Statistical Analysis 3: Comparison: Robot-assisted Therapy vs Intensive Comparison Therapy; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.81, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.54, 95% CI 2-sided [-3.87 to 4.94]
Statistical Analysis 4: Comparison: Robot-assisted Therapy vs Intensive Comparison Therapy; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 1, analysis 2]; Mean Difference (Net) = 1.19, 95% CI 2-sided [-2.74 to 5.12]

3. Secondary Outcome: Wolf Motor Function Test
Description: The Wolf Motor Function Test (WMFT) is a functionally-based test designed to provide an objective measure of both proximal (during tasks such as lifting the hand from table to box top) and distal control (grasping pencil, bringing soda can to mouth) of the paretic arm for patients after stroke or traumatic brain injury. The WMFT consists of 17 items, of which 15 measure time to perform functional tasks. The tasks are averaged to produce a score in seconds that ranges from 0 to 120 seconds, with higher scores indicating worse functioning. Outcome measure is the change in the Wolf score at 6, 12, 24 and 36 weeks relative to baseline.
Time Frame: 6, 12, 24 and 36 weeks minus baseline
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Robot-assisted Therapy | Intensive Comparison Therapy | Usual Care
Number analyzed (Participants) | 47 | 46 | 27
Seconds
  6 weeks minus baseline | -3.98 (2.72) | -3.24 (2.64) | 7.38 (2.53)
  12 week minus baseline | -3.96 (3.00) | -4.89 (3.00) | 7.54 (2.97)
  24 weeks minus baseline | -5.97 (2.77) | -3.08 (2.74) | 8.59 (3.10)
  36 weeks minus baseline | -6.23 (2.83) | -2.66 (2.79) | 7.30 (2.44)
Statistical Analysis 1: Comparison: Robot-assisted Therapy vs Usual Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.22, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; Analysis is change at 12 weeks minus baseline adjusted for the study site as a fixed effect, the Comorbidity Disease Index, and baseline WMFT value; Mean Difference (Net) = -4.41, 95% CI 2-sided [-11.52 to 2.70]
Statistical Analysis 2: Comparison: Robot-assisted Therapy vs Usual Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 1, analysis 2]; Mean Difference (Net) = -8.10, 95% CI 2-sided [-13.61 to -2.60]
Statistical Analysis 3: Comparison: Robot-assisted Therapy vs Intensive Comparison Therapy; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.82, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = 0.93, 95% CI 2-sided [-7.03 to 8.89]
Statistical Analysis 4: Comparison: Robot-assisted Therapy vs Intensive Comparison Therapy; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 1, analysis 2]; Mean Difference (Net) = -2.13, 95% CI 2-sided [-9.20 to 4.93]

4. Secondary Outcome: Change in the Numeric Rating Scale (NRS) at 12 Weeks Relative to Baseline
Description: The Numeric Rating Scale (NRS) for pain is a self report scale ranging from 0 (no Pain) to 10 (pain as bad as you can imagine).
Time Frame: 12 weeks minus baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Robot-assisted Therapy | Intensive Comparison Therapy | Usual Care
Number analyzed (Participants) | 47 | 46 | 27
units on a scale | -0.61 (0.29) | 0.24 (0.30) | 0 (0.38)
Statistical Analysis 1: Comparison: Robot-assisted Therapy vs Usual Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.08, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; Analysis of covariance at 12 weeks, adjusted for study site as a fixed effect, Comorbidity Disease Index, and the baseline value of the outcome; Mean Difference (Net) = -0.81, 95% CI 2-sided [-1.73 to 0.11]
Statistical Analysis 2: Comparison: Robot-assisted Therapy vs Intensive Comparison Therapy; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.03, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -0.84, 95% CI 2-sided [-1.62 to -0.06]

5. Secondary Outcome: Change in the Modified Ashworth Scale for Spasticity at 12 Weeks Relative to Baseline
Description: The Modified Ashworth Scale for spasticity is a measurement of spasticity across 9 muscle groups. Each muscle group is scored on a 0 to 5 scale with higher scores indicating worse functioning. The total score is the average score from the 9 muscle groups and ranges from 0 to 5 with higher scores indicating worse functioning.
Time Frame: 12 weeks minus baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Robot-assisted Therapy | Intensive Comparison Therapy | Usual Care
Number analyzed (Participants) | 47 | 46 | 27
units on a scale | -0.07 (0.09) | 0.12 (0.09) | -0.04 (0.11)
Statistical Analysis 1: Comparison: Robot-assisted Therapy vs Usual Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.95, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.25 to 0.26]
Statistical Analysis 2: Comparison: Robot-assisted Therapy vs Intensive Comparison Therapy; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.10, ANCOVA — All p-values are 2-sided with a significance level of 0.022 to adjust for multiple comparisons and interim analyses; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.42 to 0.04]

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored and collected over the entire participant follow-up period of 36 weeks
Description: Site personnel inquired about adverse and serious adverse events at each study contact.
Arm/Group | Robot-assisted Therapy | Intensive Comparison Therapy | Usual Care
Serious Adverse Events (participants affected / at risk) | 11/49 | 18/50 | 9/28
Other Adverse Events (participants affected / at risk) | 12/49 | 9/50 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robot-assisted Therapy (N=49) | Intensive Comparison Therapy (N=50) | Usual Care (N=28)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0)
Drug interaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respite care (Social circumstances) | 1 (1) | 1 (2) | 1 (2)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Colon polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Disorders (Cardiac disorders) | 1 (2) | 2 (3) | 3 (3) — Sum of all adverse event terms in the Cardiac Disorders System Organ Class
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) — Sum of all adverse event terms in the Gastrointestinal Disorders System Organ Class
General Disorders (General disorders) | 1 (1) | 2 (2) | 1 (1) — Sum of all adverse event terms in the General Disorders System Organ Class
Hepatobiliary Disorders (Hepatobiliary disorders) | 2 (4) | 0 (0) | 0 (0) — Sum of all adverse event terms in the Hepatobiliary Disorders System Organ Class
Infections (Infections and infestations) | 3 (5) | 2 (2) | 1 (1) — Sum of all adverse event terms in the Infections and Infestations System Organ Class
Injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 1 (1) — Sum of all adverse event terms in the Injury, Poisoning and Procedural Complications System Organ Class
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) — Sum of all adverse event terms in the Neoplasms System Organ Class
Nervous System Disorders (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1) — Sum of all adverse event terms in the Nervous System Disorders System Organ Class
Psychiatric Disorders (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) — Sum of all adverse event terms in the Psychiatric Disorders System Organ Class
Renal and Urinary Disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) — Sum of all adverse event terms in the Renal and Urinary Disorders System Organ Class
Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) — Sum of all adverse event terms in the Respiratory Disorders System Organ Class
Social Circumstances (Social circumstances) | 1 (1) | 1 (2) | 1 (2) — Sum of all adverse event terms in the Social Circumstances System Organ Class
Surgical and Medical Procedures (Surgical and medical procedures) | 0 (0) | 2 (2) | 2 (2) — Sum of all adverse event terms in the Surgical and Medical Procedures System Organ Class
Vascular Disorders (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) — Sum of all adverse event terms in the Vascular Disorders System Organ Class
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robot-assisted Therapy (N=49) | Intensive Comparison Therapy (N=50) | Usual Care (N=28)
Pain, Stiffness, or Soreness (General disorders) | 10 (23) | 6 (7) | 0 (0) — Only related adverse event were collected. Pain, stiffness, or soreness collected as a single type of event
Fatigue (General disorders) | 3 (6) | 0 (0) | 0 (0) — Fatigue related to study therapy.
Swelling or Bruising (General disorders) | 1 (1) | 1 (3) | 0 (0) — Swelling or Bruising collected as one event related to study therapy.
Cut, Scratch or Irritation (General disorders) | 2 (2) | 2 (2) | 0 (0) — Cut, Scratch or Irritation related to study therapy collected as one event type.
Numbness (General disorders) | 2 (2) | 0 (0) | 0 (0) — Numbness related to study therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No